CLINICAL TRIAL: NCT03815942
Title: Phase I/II Open Label Non-randomised Safety and Efficacy Study of the Viral Vectored ChAd-MVA 5T4 Vaccine in Combination With PD-1 Checkpoint Blockade in Low- or Intermediate-risk Localized or Locally Advanced Prostate Cancer and Advanced Metastatic Prostate Cancer
Brief Title: VAccination in Early and ADvanced Prostate caNCEr
Acronym: ADVANCE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: COVID stopped all trials - and ADVANCE could not restart again after the pandemic
Sponsor: University of Oxford (Other)
Collaborators: Barinthus Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADVANCE
Record Dates: First submitted 2019-01-04; First posted 2019-01-24 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Intermediate Risk Prostate Cancer; Castration-resistant Prostate Cancer
MeSH Terms: interventions — Nivolumab; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermediate risk prostate cancer (Experimental): ChAdOx1.5T4 on week 0 followed by booster injection of MVA.5T4 and nivolumab infusion on week 1. Patients will undergo radical prostatectomy on week 6.
  Interventions: Biological: ChAdOx1-MVA 5T4 vaccine; Drug: Nivolumab Infusion [Opdivo]
- Advanced metastatic prostate cancer (Experimental): ChAdOx1.5T4 on week 0 followed by booster injections of MVA.5T4 on week 4, ChAdOx1.5T4 on week 12 and MVA.5T4 on week 16. Nivolumab infusions are to be administered on week 4, 8 and 12.
  Interventions: Biological: ChAdOx1-MVA 5T4 vaccine; Drug: Nivolumab Infusion [Opdivo]

INTERVENTIONS:
Biological: ChAdOx1-MVA 5T4 vaccine — ChAdOx1.5T4 will be administered intramuscularly in an extremity (e.g. thigh) at a dose of 2.5 x10^10 virus particles followed by MVA.5T4 administered via the same route at the dose of 2x10^8 plaque forming units
Drug: Nivolumab Infusion [Opdivo] — Nivolumab is to be administered as a flat dose of 480 mg over approximately 60-minutes via IV infusion
  Other Names: anti-PD-1 monoclonal antibody

SUMMARY:
This is a clinical trial of a new treatment for prostate cancer that is a type of vaccine that could be a new way to treat cancer. A vaccine that could alert the immune system to the presence of cancer cells in the body may enable the immune system to target and kill those cells effectively. This vaccine is intended to work by making the immune system kill cells that have a special protein (called 5T4) that is present on the surface of cancer cells. The vaccine is made up of two recombinant viruses ("ChAdOx1"- chimpanzee adenovirus Ox1 and "MVA" - modified vaccinia Ankara) that have been designed to produce the 5T4 protein and have been modified so that they are weakened and cannot reproduce themselves within the body like normal viruses. Once injected into the body, these viruses make the 5T4 protein and help the body's immune system to learn to target this protein and destroy cancer cells.

This vaccine will be used in combination with the immunotherapy drug called nivolumab which is an anti-PD-1 (Programmed Death protein-1) monoclonal antibody. This is a molecule that releases the brakes on the immune system and helps the immune system to kill cancer cells more efficiently. Nivolumab as a monotherapy was approved for treatment of several tumour types but not for the prostate cancer.

This study will evaluate the safety and efficacy of ChAdOx1-MVA 5T4 vaccine in combination with nivolumab in low and intermediate risk prostate cancer patients who have elected to have their prostate removed and in patients with advanced metastatic prostate cancer.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the safety and efficacy of a combination of two new vaccines (ChAdOx1.5T4 and MVA.5T4) with a monoclonal antibody (PD-1 mAb, also known as Nivolumab and Opdivo®) against Prostate Cancer.

A vaccine that alerts the immune system to the presence of cancer cells in the body may enable the immune system to target and kill those cells effectively. This vaccine is intended to work by making the immune system kill cells that have a special protein (called 5T4) that is present on the surface of cancer cells. The use of two different forms of the vaccine has been shown to generate a more effective immune response.

ChAdOx1.5T4 consists of a virus (ChAdOx1), which is a weakened version of a chimpanzee adenovirus that has been genetically altered so that it is impossible for it to grow in humans. Modified Vaccinia virus Ankara (MVA) is licensed as third-generation vaccine against smallpox and serves as a potent vector system for development of new candidate vaccines against infectious diseases and cancer.

To both viruses we have added genes that make the 5T4 protein that is present in prostate cancer cells and which is essential to the cancer. By vaccinating, we are hoping to make the body recognise and develop an immune response to these proteins that will neutralise the effects of the cancer in human cells and therefore prevent the infection responsible for the disease.

Nivolumab (PD-1 mAb) is an immune checkpoint inhibitor. Immune checkpoints are a normal part of the immune system. Their role is to prevent an immune response from being so strong that it destroys healthy cells in the body. Immune checkpoints engage when proteins on the surface of immune cells called T cells recognize and bind to partner proteins on other cells, such as some tumour cells. These proteins are called immune checkpoint proteins. When the checkpoint and partner proteins bind together, they send an "off" signal to the T cells. This can prevent the immune system from destroying the cancer. Immunotherapy drugs called immune checkpoint inhibitors work by blocking checkpoint proteins from binding with their partner proteins. This prevents the "off" signal from being sent, allowing the T cells to kill the cancer cells. Nivolumab as a monotherapy has been approved for treatment of several tumour types but not currently for prostate cancer.

The intent was to have two cohorts of participants: Group 1 were patients who had been diagnosed with low- or intermediate-risk non-metastatic prostate adenocarcinoma and who were scheduled for radical prostatectomy; Group 2 comprised patients with metastatic castration resistant prostate cancer (mCRPC) with evidence of progression on anti-androgens.

Unfortunately, it proved impossible to recruit participants into Group 1, so the trial proceeded with just Group 2.

It was planned that the results would be measured by a composite response rate defined as one of the following:

* reduction of circulating tumour DNA of ≥50%
* serum PSA decrease of ≥50%

However, the analysis to measure the circulating tumour DNA (ctDNA) was not done for any of the participants due to the trial ending prematurely because of the COVID-19 pandemic in 2020.

The trial and the follow-up of participants was severely hampered by the Covid-19 pandemic.

In this study, we have shown that the candidate 5TA vaccines given were safe and well-tolerated. No serious adverse reactions occurred during the follow-up period. Most adverse events reported were mild or moderate in severity and all resolved spontaneously. The profile of adverse events reported in this trial is similar to other ChAdOx1 vectored vaccines.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Histologically confirmed adenocarcinoma of the prostate cancer
* Any antineoplastic therapy must have been completed a minimum of 28 days prior to enrolment
* Systemic antimicrobial therapy must have been completed a minimum of 7 days prior to enrolment
* An archival specimen of tumour tissue should be available
* Baseline laboratory parameters must meet the following criteria:

Haemoglobin ≥ 80 g/L, White cell count ≥ 2.0 x10^9/L, Neutrophils ≥ 1.5 x10^9/L, Lymphocytes ≥ 0.5 x10^9/L, Platelets ≥ 100 x10^9/L, Creatinine Clearance ≥ 40 ml/min by Cockcroft Gault formulation, Total Bilirubin ≤ 1.5 ULN, Alanine Aminotransferase ≤ 1.5 ULN, Amylase ≤ 1.5 ULN

For surgical cohort:

* Clinically localised or locally advanced disease deemed operable by the treating consultant urological surgeon i.e.: Gleason score ≤ 7, local tumour stage ≤T3c and deemed operable, no evidence of metastases (Nx/N0 and Mx/M0), no evidence of high grade Gleason 5 disease, PSA ≤ 20 ng/ml
* Scheduled for and considered fit for radical prostatectomy

For advanced metastatic cohort:

* Evidence of at least one distant metastasis based on MRI, CT, PET or bone scintigraphy
* Established on and suitable to continue with androgen deprivation therapy (ADT) using any luteinizing hormone releasing hormone (LHRH) agonist
* On treatment with anti-androgen therapy using either abiraterone (Zytiga®) or enzalutamide (Xtandi®) and demonstrating evidence of disease progression at the time of enrolment
* Suitable to continue therapy with either abiraterone or enzalutamide at the time of enrolment at discretion of their managing clinician
* Patients who have received chemotherapy following progression on androgen-targeting therapies are eligible
* Satisfactory functional status defined as ECOG Performance Status ≤ 1

Exclusion Criteria:

For all participants:

* Any prior diagnosis or clinical suspicion of autoimmune disease
* History of allergic disease or reaction likely to be exacerbated by any component of the vaccine, e.g. egg products
* Other prior malignancy with an estimated ≥ 30% chance of relapse within 2 years
* Participation in another research study involving an investigational product or investigational surgical procedure in the 30 days preceding enrolment, or planned use during the study period
* Any prior exposure to checkpoint inhibitor drugs including anti-PD-1, anti-PD-L1, or anti-CTLA-4 monoclonal antibodies or any prior treatment with investigational vaccines
* Administration of immunoglobulins and/or any blood products within the one month preceding the planned administration of the study drugs
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Any confirmed or suspected immunocompromised state
* Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema
* History of anaphylaxis in relation to vaccination or any clinically significant allergic disease likely to be exacerbated by any component of the vaccine or checkpoint inhibitor preparations

For advanced metastatic cohort:

* The treating oncologist estimates a subject's life expectancy to be ≤ 6 months
* Any active, previously treated, or suspected intracranial or leptomeningeal metastases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, Study Director — University of Oxford; Freddie Hamdy, Study Director — Nuffield Department of Surgical Sciences, Oxford University Hospitals NHS Foundation Trust; Andrew Protheroe, Principal Investigator — Nuffield Department of Surgical Sciences, Oxford University Hospitals NHS Foundation Trust; Peter Hoskin, Principal Investigator — Department of Oncology, The Christie NHS Foundation Trust; Mark Tuthill, Study Chair — Oxford Cancer and Haematology Centre, Oxford University Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Department of Oncology, The Christie NHS Foundation Trust, Manchester
  - Cancer and Haematology Centre, Churchill Hospital, Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No
The results in anonymised summary will be shared in publications resulting from the trial.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intermediate Risk Prostate Cancer | Advanced Metastatic Prostate Cancer
Started | 0 (This arm was not able to recruit any participants - so did not happen.) | 23
Completed | 0 (Unable to recruit any participants) | 6
Not Completed | 0 | 17
Not completed — Withdrawal by Subject | 0 | 17

BASELINE CHARACTERISTICS:
Population: No participants were recruited to the Intermediate risk prostate cancer arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Intermediate Risk Prostate Cancer | Advanced Metastatic Prostate Cancer | Total
Number analyzed (Participants) | 0 | 23 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 0 | 21 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 23 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom |  | 23 | 23
Serum PSA [Number; unit: participants] — Participants whose Serum PSA baseline was measured
  participants |  | 23 | 23

OUTCOME MEASURES:

1. Primary Outcome: Safety - Incidence of Treatment-related Adverse Events.
Description: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0.
  Note: All participants had one or more adverse events during the period they were monitored.
Time Frame: From baseline to 12 months
Population: No participants were recruited in the Intermediate risk prostate cancer group
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate Risk Prostate Cancer | Advanced Metastatic Prostate Cancer
Number analyzed (Participants) | 0 | 23
Participants |  | 23

2. Primary Outcome: Efficacy - Measure Composite Response Rate Defined as One of the Following: 1) Change in Circulating Tumour DNA 2) Change in Serum PSA
Description: Evaluate the efficacy by assessing the number of participants with 50% or more change in ctDNA or PSA concentration in the blood from baseline to 12 months post treatment.
  Change in serum PSA was analysed for this outcome as one the two alternative methods planned.
  As described in the trial overview, no ctDNA analysis was done due to the trial closing prematurely because of COVID-19 - by the time the pandemic had finished, the facility to perform the ctDNA analysis option was no longer available. Because no laboratory analysis was done, there is no data to report.
Time Frame: From baseline to 12 months
Population: No participants recruited to the Intermediate risk prostate cancer arm. Change in serum PSA was analysed for this outcome as one the two alternative methods planned.
  As described in the trial overview, no ctDNA analysis was done due to the trial closing prematurely because of COVID-19 - by the time the pandemic had finished, the facility to perform the ctDNA analysis option was no longer available.
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate Risk Prostate Cancer | Advanced Metastatic Prostate Cancer
Number analyzed (Participants) | 0 | 23
Participants |  | 5

3. Secondary Outcome: Evaluate Immune Responses to the Vaccine Antigen in the Periphery
Description: Number of participants with peripheral 5T4-specific T cell responses secondary to treatment
Time Frame: From baseline to 12 months
Population: No participants recruited to the Intermediate risk prostate cancer arm
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate Risk Prostate Cancer | Advanced Metastatic Prostate Cancer
Number analyzed (Participants) | 0 | 23
Participants |  | 23

4. Secondary Outcome: Evaluate Immune Cell Subsets in the Prostate Secondary to Treatment (for Surgical Cohort)
Description: Number of participants with intraprostatic infiltration of CD3+CD8+ T cells secondary to treatment
Time Frame: From baseline to radical prostatectomy, an expected average of 6 weeks
Population: No participants recruited to the Intermediate risk prostate cancer arm
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate Risk Prostate Cancer | Advanced Metastatic Prostate Cancer
Number analyzed (Participants) | 0 | 23
Participants |  | 23

5. Secondary Outcome: Evaluate Progression-free Survival Following Study Treatment (for Advanced Metastatic Cancer Cohort)
Description: Evaluating the number of participants experiencing progression-free survival at 6 and 12 months post treatment
Time Frame: 6-12 months
Population: No participants recruited to the Intermediate risk prostate cancer arm
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate Risk Prostate Cancer | Advanced Metastatic Prostate Cancer
Number analyzed (Participants) | 0 | 23
Participants |  | 23

6. Secondary Outcome: Evaluate Overall Survival Following Study Treatment (for Advanced Metastatic Cancer Cohort)
Description: Evaluating the number of participants experiencing overall survival at 6 and 12 months post treatment
Time Frame: 6-12 months
Population: No participants recruited to the Intermediate risk prostate cancer arm
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate Risk Prostate Cancer | Advanced Metastatic Prostate Cancer
Number analyzed (Participants) | 0 | 23
Participants |  | 23

ADVERSE EVENTS:
Time Frame: For 12 months following study treatment. Note that a number of participants withdrew from the study before the 12 months had elapsed.
Description: Assessment of serious events was performed according to ICH-GCP guidelines.
Arm/Group | Intermediate Risk Prostate Cancer | Advanced Metastatic Prostate Cancer
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/0 | 9/23
Other Adverse Events (participants affected / at risk) | 0/0 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermediate Risk Prostate Cancer (N=0) | Advanced Metastatic Prostate Cancer (N=23)
fatigue/haematura/increasing lymphoedema (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Possibly urosepsis (Renal and urinary disorders) | 0 (0) | 1 (1)
Worsening renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Metastatic spinal cord compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
increasing back pain & right arm weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pyrexia and rigors (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
progressive lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Suspected pulmonary clots -> Chest infection (lifelong smoker) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermediate Risk Prostate Cancer (N=0) | Advanced Metastatic Prostate Cancer (N=23)
Fatigue (General disorders) | 0 (0) | 22 (22)
Fever (General disorders) | 0 (0) | 7 (7)
Headache (General disorders) | 0 (0) | 2 (2)
Myalgia (General disorders) | 0 (0) | 10 (10)
Arthralgia (General disorders) | 0 (0) | 7 (7)
Anorexia (General disorders) | 0 (0) | 9 (9)
Rash (General disorders) | 0 (0) | 10 (10)
Itch General (General disorders) | 0 (0) | 2 (2)
Itch (Local) (General disorders) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Abdominal pain (General disorders) | 0 (0) | 7 (7)
Urinary (Renal and urinary disorders) | 0 (0) | 10 (10)
Warmth (General disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 4 (4) — including indigestion and "Lower abdominal discomfort"
acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Altered sensation right finger/thumb (Nervous system disorders) | 0 (0) | 3 (3) — including "Middle finger nerve changes" and "Peripheral neuropathy"
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (3) — including Fatigue
Back ache (General disorders) | 0 (0) | 6 (6) — or back pain including "Lower back pain" and "Occasional back ache"
Bilateral lower limb oedema (Blood and lymphatic system disorders) | 0 (0) | 3 (3) — including Lymphoedema
Bilateral Subconjunctival Ulcers (Eye disorders) | 0 (0) | 2 (2) — including "subconjunctival ulcers"
Black stools (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloatedness (General disorders) | 0 (0) | 1 (1)
Breathlessness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — including Dyspnoea
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Chest infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) — including "cold" and "flu" and "Lower respiratory tract infection"
Collapse (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 7 (7)
Diarrhoea and vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) — including Faecal Urgency
Discomfort (right) sacrum (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (7) — Including "Hip Pain" either side and "Pain Bilateral Buttocks" and "Pain left buttock" and "Pain right hip"
Dizziness (General disorders) | 0 (0) | 1 (1)
Dry mouth (General disorders) | 0 (0) | 2 (2)
Elevated Amylase (Investigations) | 0 (0) | 1 (1)
Fall (General disorders) | 0 (0) | 2 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hot flushes (General disorders) | 0 (0) | 1 (1)
Hypercalcemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperglycemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
hypotension post vaccine (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — including Low BP diastolic
Kidney function (Renal and urinary disorders) | 0 (0) | 1 (1)
left thigh wart (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Leg Ache / weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (8) — includes "Occasional left calf pain" and "Pain in knees" and "Pain left calf" and "Stiff leg" and "Thigh Pain" and "Weakness right leg"
Lack of appetite (General disorders) | 0 (0) | 1 (1)
Low mood (General disorders) | 0 (0) | 1 (1)
Lower abdomen skin lesions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
lymphocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 0 (0) | 1 (2)
pain in arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pain injection site L thigh (General disorders) | 0 (0) | 2 (3) — including "Tender injection site"
PR Bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Raised ALT (Hepatobiliary disorders) | 0 (0) | 1 (1)
Raised temperature (General disorders) | 0 (0) | 1 (1)
rash right leg and hand (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rib pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right Iliac pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Shivery (General disorders) | 0 (0) | 1 (1)
Sore mouth (General disorders) | 0 (0) | 3 (3) — including "sore throat"
Stiff joints (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stye left lower eyelid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 2 (2)
thrombosis in the coeliac axis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Tooth Ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) — including "tooth abscess"
Vertigo (General disorders) | 0 (0) | 1 (1)
Lethargy (General disorders) | 0 (0) | 1 (1)
Buttock abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial finished prematurely due to the COVID-19 pandemic in 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT03815942/Prot_000.pdf